CLINICAL TRIAL: NCT03289689
Title: The Acute Effects of Whole-Body Vibration on Manual Ability Performance: A Randomized Controlled Trial
Brief Title: Whole-body Vibration and Manual Ability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URJC
Record Dates: First submitted 2017-07-13; First posted 2017-09-21 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Body Weight; Vibration; Motor Activity
MeSH Terms: conditions — Body Weight; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration (Experimental): The subjects in the WBV group performed one series of five consecutive repetitions of 60 sec unsynchronised multidimensional WBV (Zeptoring, Scisen GmbH, Germany; 4 Hz, amplitude 3mm) with a 1-min pause between administrations, three times a week. The construction of this device is designed to perform a nonharmonious generation of oscillating movements in vertical and horizontal planes in order to prevent occurrences of resonance and habituation of receptors.
  During the intervention, subjects wore thin-soled gymnastic-type shoes, carrying out in a squatting standing position, with slight flexion at the hips, knees and ankle joint, on the vibration platform.
  Interventions: Device: Whole-body vibration (WBV)
- Control (No Intervention): The controls did not receive any training.

INTERVENTIONS:
Device: Whole-body vibration (WBV) — Whole-body vibration (WBV) is a novel neuromuscular therapeutic intervention that has recently been developed since in the mid-1960s. Hagbart and Eklund showed in human experiments that a reflex muscle contraction can result as a consequence of applying vibrations to the muscular-tendon system. The subjects stand on a platform that generates stochastic vibrations at a frequency between 1-12.5 Hz.
  Arms: Whole body vibration

SUMMARY:
Purpose: To evaluate the short-term effects of whole-body vibration (WBV), using reciprocating plate technique, on manual ability performance in healthy younger.

Material and methods: 38 healthy young volunteers were randomized to WBV group (N=19; 6 men, 13 women; mean age 21, 3.8yrs) or control group (N=19; 6 men, 13 women; mean age 20.5, 3.5yrs). The subjects in the WBV group performed one series of five consecutive repetitions of 60 sec unsynchronised WBV (Zeptoring, Scisen GmbH, Germany; 4 Hz, amplitude 3mm) with a 1-min pause between administrations, three times a week. The controls did not receive any training. Both groups were evaluated at baseline and after intervention, in the Rey Juan Carlos University´s Gait Analysis Laboratory. Four outcome measures of Purdue Pegboard test (PPT): preferred hand (PH), non-preferred hand (NPH), both hands (BH) and assembly (A) was performed baseline and 5 min after intervention.

ELIGIBILITY:
Inclusion criteria:

- Healthy subjects aged between 18 and 30 years.

Exclusion criteria:

* Contraindication for WBV: pregnancy, recent fractures, malignancies, kidney stones, cardiac pacemaker, infectious disease or recent thromboembolic.
* Subjects with any musculoskeletal o neurological disorders that affected their hands.
* Individuals already treated with WBV were excluded.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-10 (Actual)

PRIMARY OUTCOMES:
Purdue Pegboard test (change) | Baseline, immediately after intervention and one month after the intervention
  Change in Purdue Pegboard test. This tool evaluates the fine dexterity

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alguacil Diego IM, Martinez Piedrola RM, Aguilera Rubio A, Gomez Alguacil M, Molina Rueda F. Acute Effects of a Week of Stochastic-Random Whole-Body Vibration on Manual Ability Performance in Healthy Subjects: A Preliminary Pilot Study. Biomed Res Int. 2025 Sep 23;2025:7662370. doi: 10.1155/bmri/7662370. eCollection 2025. PMID 41031241